CLINICAL TRIAL: NCT06146790
Title: Evaluation of Endovascular Treatment in Acute Intracranial Distal Medium Vessel Occlusion Stroke - a Multicenter, Randomized Controlled, Clinical Trial
Brief Title: Evaluation of Endovascular Treatment in Acute Intracranial Distal Medium Vessel Occlusion Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Wei Hu, Professor, The First Affiliated Hospital of University of Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORIENTAL-MeVO
Record Dates: First submitted 2023-11-10; First posted 2023-11-27 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Acute Ischemic Stroke; Endovascular Thrombectomy
Keywords: Medium Vessel Occlusion; Stroke Due To Medium Vessel Occlusion; Endovascular Treatment; Standard Medical Management
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular treatment+ standard medical management (Experimental): For the subjects randomized to endovascular treatment (EVT), treatment initiation is defined as the date and time of arterial puncture. Ideally, femoral artery puncture will occur within 30 minutes of randomization and no longer than 60 minutes after the completion of the qualifying imaging. Treatment initiation (arterial puncture) must occur before 24 hours since the subject was last known well. Date and time of arterial puncture, revascularization, and procedure end will be recorded. It is expected that the interventional procedure will be completed within two (2) hours of arterial access. If an appropriate thrombus or residual stenosis is identified, the choice of EVT strategy will be made by the treating neurointerventionalist. All mechanical thrombectomy devices for EVT, which are approved by CFDA for this purpose, are allowed in the trial.
  Interventions: Procedure: endovascular treatment
- Standard medical management (Active Comparator): Standard medical management
  Interventions: Other: Standard medical management

INTERVENTIONS:
Procedure: endovascular treatment — For the subjects randomized to endovascular treatment (EVT) treatment initiation is defined as the date and time of arterial puncture. Ideally, femoral artery puncture will occur within 30 minutes of randomization and no longer than 60 minutes after the completion of the qualifying imaging. Treatment initiation (arterial puncture) must occur before 24 hours since the subject was last known well.Date and time of arterial puncture, revascularization, and procedure end will be recorded. It is expected that the interventional procedure will be completed within two (2) hours of arterial access. If an appropriate thrombus or residual stenosis is identified, the choice of EVT strategy will be made by the treating neurointerventionalist. All mechanical thrombectomy devices for EVT, which are approved by CFDA for this purpose, are allowed in the trial.
  Arms: Endovascular treatment+ standard medical management
Other: Standard medical management — Standard medical management
  Arms: Standard medical management

SUMMARY:
Rationale: Distal Medium Vessel Occlusion (MeVO) are thought to cause as many as 25% to 40% of all acute ischemic strokes (AIS). Despite their relatively high frequency, there is no consensus regarding the optimal management of these patients. However, the fact that AIS related to MeVO often results in significant disability despite best medical treatment (including intravenous thrombolysis, IVT) calls for novel treatment approaches. Fortunately, a growing number of non-randomized studies have now been published demonstrating the feasibility of endovascular treatment (EVT) for MeVO strokes. These studies have demonstrated that distal EVT leads to high rates of successful reperfusion and may be performed with a comparable safety profile to that of EVT for proximal arterial occlusions. Therefore, a strong rational exists to test the safety and efficacy of EVT for MeVO stokes in a prospective randomized clinical trial.

Objectives: The primary objective of this study is to evaluate the hypothesis that endovascular thrombectomy is superior to standard medical management in achieving more favorable outcomes according to the modified Rankin Scale scores at 90 days in subjects presenting with acute ischemic stroke related to a distal medium vessel occlusion within 24 hours from symptom onset (defined as time last know well, TLKW).

Secondary objectives include the assessment of the cost-effectiveness of endovascular thrombectomy in the medium vessel occlusion (MeVO) population as well as its impact on health-related quality of life.

Study design: The study is a prospective, multicenter, investigational, randomized, controlled, open-label study with blinded endpoint evaluation (PROBE design) and an adaptive design with population enrichment.

Study population: Subjects presenting with acute ischemic stroke within 24 hours from TLKW and whose strokes are attributable to a distal medium vascular occlusion defined as co/non-dominant M2 segment or M3 segment of the MCA, the ACA (A1, A2, or A3 segments), or the PCA (P1, P2 or P3 segments) with evidence of salvageable brain tissue on perfusion imaging, M2 segment vessel diameter should not exceed 2.0 mm.

Primary outcome: Shift in distribution of all levels of the 90-day the modified Rankin Scale with levels 5-6 combined (mRS; 0, 1, 2, 3, 4, 5-6) as assessed by structured assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years (no upper age limit).
2. Evidence of a primary (e.g., not secondary to EVT of proximal vessel occlusion) distal medium vascular occlusion defined as occlusion of the co/non-dominant M2 segment* or M3 segment of the MCA, the ACA (A1, A2, or A3 segments), or the PCA (P1, P2 or P3 segments) resulting in significant clinical deficits and expected to be treatable by endovascular thrombectomy.

   * Co/non-dominant M2 segment vessel diameter should not exceed 2.0 mm. Co-dominant supplying 50% of the MCA territory vs non-dominant supplying <50% of the MCA territory.
3. Premorbid mRS ≤ 2.
4. Baseline National Institutes of Health Stroke Scale (NIHSS) score ≥6 at the time of randomization.
5. Time from onset (or time last seen well) to randomization<24 hours.
6. For patients with more than 6 hours of onset (or time last seen well), Clinical-Imaging mismatch assessment defined as any of the following scenarios (A or B):

   A. Non-contrast CT of the head or Brain MRI DWI lesion with <50% involvement of the vascular territory corresponding to the clinical manifestation:

   B. Target Mismatch Profile on CT perfusion or MRI (Mismatch Volume >10cc and mismatch Ratio >1.4 ).
7. Informed consent obtained from patient or acceptable patient surrogate.

Exclusion Criteria:

1. Any sign of intracranial hemorrhage on baseline CT/MR (SDH/SAH/ICH).
2. Rapidly improving symptoms, particularly if in the judgment of the managing clinician that the improvement is likely to result in the patient having an NIHSS score of <6 at randomization.
3. Significant ischemic changes in a territory other than the occluded site that in the opinion of the investigator could reduce the benefit of endovascular treatment.
4. Contra indication to imaging with MR or CT with contrast agents.
5. Any terminal illness such that patient would not be expected to survive more than 1 year.
6. Recent past history or clinical presentation of ICH, subarachnoid hemorrhage (SAH), arterio-venous (AV) malformation, aneurysm, or cerebral neoplasm other than meningioma.
7. Any imaging findings suggestive of futile recanalization in the judgment of the local investigator.
8. seizures at stroke onset if it precludes obtaining an accurate baseline NIHSS.
9. Baseline blood glucose of <50 mg/dL (2.78 mmol) or >400 mg/dL (22.20 mmol).
10. Known history of hereditary or acquired hemorrhagic diathesis and/or platelet count <50×109/L.
11. Known renal failure as defined as serum creatinine levels > 260umol/l（3.0 mg/dL）.
12. Presumed septic embolus or suspicion of bacterial endocarditis.
13. Any other condition that, in the opinion of the investigator could impose hazards to the patient or affect the participation of the patient in the study if an endovascular procedure was performed.
14. History of drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
15. Subjects with occlusions in multiple vascular territories (e.g., bilateral or multi-territorial anterior circulation, or anterior/posterior circulation)
16. Subject participating in a study involving an investigational drug or device that would impact this study.
17. Known pregnancy.
18. Prisoner or incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The 90-day modified Rankin Scale (mRS) | 90 (± 14 days) after procedure
  Shift in distribution of all levels of the 90-day modified Rankin Scale with levels 5-6 combined (mRS; 0, 1, 2, 3, 4, 5-6) as assessed by structured assessment.

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | 90 (± 14 days) after procedure
  Shift in distribution of the 90-day mRS (0;1;2;3;4;5;6) as assessed by structured assessment.
Independent Outcome | 90 (± 14 days) after procedure
  Rates of Independent Outcome defined as mRS ≤2 and/ or equal to Baseline mRS at 90 days
Excellent Outcome | 90 (± 14 days) after procedure
  Rates of Excellent Outcome defined as mRS ≤1 and/ or equal to Baseline mRS at 90 days
Good Functional Outcomes | 90 (± 14 days) after procedure
  Rates of Good Functional Outcomes adjusted for the baseline mRS and stroke severity (NIHSS) according to the modified Rankin Scale scores at 90 days as following:
  * If NIHSS <10 and Baseline mRS 0 or 1: 90-day mRS ≤1
  * If NIHSS <10 and Baseline mRS 2: 90-day mRS ≤2
  * If NIHSS ≥10 and Baseline mRS 0 or 1: 90-day mRS ≤2
  * If NIHSS ≥10 and Baseline mRS 2: 90-day mRS ≤3

OTHER OUTCOMES:
Mortality | 90 (± 14 days) after procedure
  Number of subjects who died at 90-day follow-up/total number of subjects who participated in 90-day follow-up) x100%
Symptomatic intracranial hemorrhage (SICH) | 24 hours (-2/+12H) after procedure
  SICH means any hemorrhage with neurological deterioration, as indicated by an NIHSS score that was higher by ≥4 points than the value at baseline or the lowest value in the first 24 hours (-2/+12) , or any hemorrhage leading to death.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, MD, PhD, Study Chair — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jing X, Nogueira RG, Nguyen TN, Tao C, Zhu Y, Li R, Sun J, Wang L, Zhang C, Liu T, Song J, Saver JL, Hu W. Endovascular treatment in acute intracranial distal medium vessel occlusion stroke: Study protocol and rationale. Int J Stroke. 2025 Jul;20(6):763-768. doi: 10.1177/17474930251332753. Epub 2025 Mar 25. PMID 40134089